CLINICAL TRIAL: NCT03289286
Title: Pilot Study Evaluating a Perioperative E-follow-up Protocol in Patients With Ambulatory Surgery for Breast Cancer
Acronym: PITCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 17SEIN04
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Ambulatory surgery; Electronic tool; e-follow-up
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with breast cancer operated in ambulatory (Other)
  Interventions: Other: Dedicated and coordinated e-follow-up.

INTERVENTIONS:
Other: Dedicated and coordinated e-follow-up. — In pre- and post-surgery:
  * Completion of questionnaires using an electronic tool,
  * Telephone follow-up if necessary between the nurse and the patient.

SUMMARY:
This is a monocentric, prospective cohort study evaluating the feasibility of a perioperative e-follow-up protocol in patients with ambulatory surgery for breast cancer.

This protocol will be based on:

* A coordinated ambulatory follow-up performed by a dedicated nurse
* An electronic follow-up tool used in pre- and post-surgery

Patients will be followed 8 days before the surgery until 30 days after the surgery of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for an ambulatory surgery of breast cancer (partial mastectomy with or without lymph node sampling)
2. Ambulatory surgery planned 10 days or more after inclusion date
3. Age > or = 18 years old
4. Affiliated to the french social security system
5. Patient must provide written informed consent prior to any study-specific procedure or assessment

Exclusion Criteria:

1. Surgery other than breast cancer surgery in ambulatory (benign breast surgery, other surgical specialities)
2. Patient who cannot connect to the electronic tool at home (no computer, no tablet computer or no internet connection)
3. Pregnant or breastfeeding women
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
5. Patient protected by law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Rate of patients without failure to the e-follow-up. A failure is defined by absence of connection to the electronic tool and the mismatch between the alert level and severity of complications. | 1.5 months by patient

SECONDARY OUTCOMES:
Patient satisfaction to the e-follow-up. | 1.5 months by patient
  Satisfaction will be evaluated by questionnaire.
The rate of patients who discontinue the study 8 days before the surgery. | 1.5 months by patient
The number of unplanned visits into the Center after ambulatory surgery in the first 24 hours and during the first 30 days will be assessed for each patient. | 1.5 months by patient
Rate of patients with at least one unplanned visit. | 1.5 months by patient
The time spent by the dedicated nurse for the follow-up protocol management. | 1.5 months by patient
  It will be defined as the sum of the time spent at different stages: initial training of patients, tracking of the connections to the tool, tracking of the alerts and telephone contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri GANGLOFF, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud IUCT-ONCOPOLE, Toulouse, France